CLINICAL TRIAL: NCT03171493
Title: Neoadjuvant Intravesical NIS Measles Virus (MV-NIS) in Patients Undergoing Cystectomy for Urothelial Carcinoma But Ineligible for Neoadjuvant Cisplatin-based Chemotherapy
Brief Title: Trial of Intravesical Measles Virotherapy in Patients With Bladder Cancer Who Are Undergoing Radical Cystectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vyriad, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VYR-MV1-102
Record Dates: First submitted 2017-03-24; First posted 2017-05-31 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: Urothelial Carcinoma
Keywords: Bladder cancer; TURBT; Radical cystectomy; BCG; Muscle Invasive Bladder Cancer; Intravesical; chemotherapy for bladder cancer; Oncolytic
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravesical MV-NIS therapy prior to radical cystectomy (Experimental): MV-NIS will be administered via intravesical instillation as a single dose on Day 1 (7, 14, 21 or 28 days before cystectomy) or two doses on Day 1 and 15 (14 and 28 days before cystectomy).
  Interventions: Biological: MV-NIS

INTERVENTIONS:
Biological: MV-NIS — Attenuated measles virus encoding NIS (MV-NIS)

SUMMARY:
This is a Phase 1 study designed to test the tolerability and feasibility of intravesical therapy with an attenuated Measles virus (MV-NIS) in patients with urothelial carcinoma who are undergoing radical cystectomy but are ineligible or do not desire neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Study VYR-MV1-102 is a Phase 1 study designed to determine the tolerability, feasibility and preliminary efficacy of attenuated MV-NIS virus after neoadjuvant intravesical administration prior to RC in patients with UC who are ineligible for current neoadjuvant chemotherapy.

Investigators will use a novel adaptive trial design that varies the time between TURBT, virus administration and RC.

Currently, intravesical administration of BCG is delayed four to six weeks after TURBT to reduce the likelihood of systemic BCG absorption and BCG sepsis. Given this clinical safety precedent, Investigators propose initial patients be treated within one week of RC to maximize the time between TURBT and MV-NIS administration.

Subsequent patients will be treated earlier before RC (up to 29 days prior), thereby reducing the interval between TURBT and virus administration to maximize the treatment duration before RC. An expansion cohort will also be used to test the feasibility, tolerability and efficacy of two repeat MV-NIS doses prior to RC. MV-NIS has been proven safe at a dose of 1x1011 TCID50 intravenously in patients lacking MV immunity (Russell 2014), which allays concern for systemic toxicity after intravesical administration even if post-TURBT administration results in systemic MV-NIS absorption.

Pathologic downstaging and CR (assessed by T0 rate) at surgery are secondary endpoints, designed to give an early indication of efficacy potential. This will facilitate future virotherapy strategies targeting replicative tumor destruction and stimulation of systemic anti-tumor immunity as possible strategies for neoadjuvant and bladder-sparing therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Urothelial carcinoma (UC) of the bladder, with histologic confirmation of primary UC pathology; indication for Radical cystectomy (RC); ineligibility for platinum-based neoadjuvant chemotherapy
* ECOG Performance Status (PS) 0 or 1.
* Ability to provide informed consent.
* Willingness to comply with all required protocol procedures including providing biologic specimens and returning to the clinical study site for follow up visits.
* Performance status sufficient to undergo RC (in the opinion of the enrolling urologist) including adequate hematological, liver and kidney function
* Must be willing to implement contraception throughout study and for 30 days following RC.

Exclusion Criteria:

* Variant UC pathology including but not limited to micropapillary, signet ring,sarcomatoid, and clear cell variants.
* Patients with any other prior malignancy are not allowed except for the following: History of or concurrent non-invasive UC involving a portion of urinary tract outside of the bladder; Adequately treated basal cell or squamous cell skin cancer; In situ cervical cancer; Adequately treated Stage I or II cancer from which the patient is currently incomplete remission or other cancer from which the patient has been disease-free for 2 years.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Any of the following prior therapy: Chemotherapy ≤ 3 weeks prior to registration. Biologic therapy ≤ 4 weeks prior to registration. Radiation therapy ≤ 3 weeks prior to registration
* Other concurrent investigational therapy (utilized for a non-FDA-approved indication and in the context of a research investigation).
* Pregnant women.
* Nursing women.
* Men or women of childbearing potential who are unwilling to employ adequate contraception during treatment and 8 weeks following the completion of study drug treatment.
* Allergy to measles vaccine or history of severe reaction to prior measles vaccination.
* History of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with intravesical MV-NIS treatment related adverse events (NCI CTCAE; Version 4.03) | 30 days after cystectomy
  Assessment of safety and toxicity of intravesical MV-NIS administration in patients with Urothelial Carcinoma undergoing cystectomy

SECONDARY OUTCOMES:
Pathologic staging at time of cystectomy following intravesical MV-NIS therapy | Measured in bladder specimen following cystectomy (up to 29 days following MV-NIS administration)
  Preliminary assessment of antitumor efficacy of intravesical MV-NIS therapy
pT0 rate at time of cystectomy following intravesical MV-NIS therapy | Measured in bladder specimen following cystectomy (up to 29 days following MV-NIS administration)
  Preliminary assessment of antitumor efficacy of intravesical MV-NIS therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bexon, MD, Study Director — CMO - Medical Monitor
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - Ochsner Health, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No